CLINICAL TRIAL: NCT01259323
Title: A Randomized, Double-Blind, Placebo-Controlled, Sequential Ascending, Repeated-Dose Study of the Safety and Pharmacokinetics of Subcutaneous REGN668 in Patients With Moderate-to-Severe Extrinsic Atopic Dermatitis
Brief Title: Sequential Ascending Dose Study to Assess the Safety and Tolerability of REGN668 (SAR231893) in Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R668-AD-0914
Record Dates: First submitted 2010-12-10; First posted 2010-12-14 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Dermatitis
MeSH Terms: conditions — Dermatitis | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental)
  Interventions: Biological: REGN668
- Cohort 2 (Experimental)
  Interventions: Biological: REGN668
- Cohort 3 (Experimental)
  Interventions: Biological: REGN668

INTERVENTIONS:
Biological: REGN668 — Dose 1: REGN668 or placebo
  Arms: Cohort 1
Biological: REGN668 — Dose 2: REGN668 or placebo
  Arms: Cohort 2
Biological: REGN668 — Dose 3: REGN668 or placebo
  Arms: Cohort 3

SUMMARY:
The purpose of this study is to assess the Safety and Tolerability of REGN668 (how the body reacts to the drug) compared to placebo (an inert substance) in patients with moderate-to-severe extrinsic Atopic Dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of atopic dermatitis that has been present for at least 3 years before the screening visit
* Investigator's Global Assessment (IGA) score of >/= 3 at the screening and baseline visits
* >/= 15% body surface area (BSA) of AD involvement at the screening and baseline visits
* History of inadequate response to a stable (>/= 1 month) regimen of topical corticosteroids or calcineurin inhibitors as treatment for AD within 3 months before the screening visit
* Willing and able to comply with clinic visits and study-related procedures
* Patient able to read and understand, and willing to sign the informed consent form

Exclusion Criteria:

* A positive QuantiFERON® - TB (tuberculosis) Gold Test at the screening visit
* Known history of Human Immunodeficiency Virus (HIV), Hepatitis B or Hepatitis C and/or positive Hepatitis B surface antigen (HBsAg), positive Hepatitis C antibody (HCV)
* Treatment with an investigational drug within 8 weeks before the baseline visit
* Treatment with leukotriene inhibitors within 4 weeks before the baseline visit
* Treatment with systemic corticosteroids within 4 weeks before the baseline visit
* Treatment with topical corticosteroids, tacrolimus, and/or pimecrolimus within 1 week before the baseline visit
* Systemic treatment for AD with an immunosuppressive/immunomodulating substance within 4 weeks before the baseline visit
* Chronic or acute infection requiring treatment
* History of clinical parasite infection, other than treated trichomoniasis
* History of malignancy within 5 years before the baseline visit
* Any medical or psychiatric condition which, in the opinion of the investigator or the sponsor's medical monitor, would place the patient at risk, interfere with participation in the study, or interfere with the interpretation of study results
* Pregnant or breast-feeding women
* Unwilling to use adequate birth control, if of reproductive potential and sexually active

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoint in the study is the incidence of treatment-emergent adverse events (TEAEs) in patients treated with REGN668 or Placebo from baseline through week 12. | 12 weeks

SECONDARY OUTCOMES:
The secondary endpoint is to characterize PK profile of study drug REGN668 from baseline through week 12. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (10):
- United States (10):
  - Los Angeles, California
  - Riverside, California
  - Miami, Florida
  - Chicago, Illinois
  - Troy, Michigan
  - New York, New York
  - Rochester, New York
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Dallas, Texas

REFERENCES:
- [Derived] Hamilton JD, Suarez-Farinas M, Dhingra N, Cardinale I, Li X, Kostic A, Ming JE, Radin AR, Krueger JG, Graham N, Yancopoulos GD, Pirozzi G, Guttman-Yassky E. Dupilumab improves the molecular signature in skin of patients with moderate-to-severe atopic dermatitis. J Allergy Clin Immunol. 2014 Dec;134(6):1293-1300. doi: 10.1016/j.jaci.2014.10.013. PMID 25482871
- [Derived] Beck LA, Thaci D, Hamilton JD, Graham NM, Bieber T, Rocklin R, Ming JE, Ren H, Kao R, Simpson E, Ardeleanu M, Weinstein SP, Pirozzi G, Guttman-Yassky E, Suarez-Farinas M, Hager MD, Stahl N, Yancopoulos GD, Radin AR. Dupilumab treatment in adults with moderate-to-severe atopic dermatitis. N Engl J Med. 2014 Jul 10;371(2):130-9. doi: 10.1056/NEJMoa1314768. PMID 25006719